CLINICAL TRIAL: NCT03748251
Title: Demystifying the Pizza Bolus: the Effect of Dough Fermentation Time on Glycemic Response in Children With Type 1 Diabetes Mellitus Receiving Sensor-augmented Pump Therapy
Brief Title: Management of Glycemia Following a Pizza Meal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Campania Luigi Vanvitelli (Other)
Collaborators: Federico II University (Other)
Responsible Party: Principal Investigator, Angela Zanfardino, Principal Investigator, University of Campania Luigi Vanvitelli
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: PZ_2018
Record Dates: First submitted 2018-11-16; First posted 2018-11-20 (Actual); Last update posted 2018-11-20 (Actual); Status verified 2018-11

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Continuous Subcutaneous Insulin Infusion; diet; postprandial glucose; postprandial hypoglycemia; postprandial hyperglycemia
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hypoglycemia; Hyperglycemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Short fermented pizza (Experimental): the patients ate a pizza that fermented for 8 hours
  Interventions: Other: the patients ate a pizza that fermented for 8 hours
- Long fermented pizza (Experimental): the patients ate a pizza that fermented for 24 hours
  Interventions: Other: the patients ate a pizza that fermented for 24 hours

INTERVENTIONS:
Other: the patients ate a pizza that fermented for 8 hours — Patients eat pizza prepared with controlled ingredients but fermented 8 hours
  Arms: Short fermented pizza
Other: the patients ate a pizza that fermented for 24 hours — Patients eat pizza prepared with controlled ingredients but fermented 24 hours
  Arms: Long fermented pizza

SUMMARY:
Glycemia following pizza consumption is typically managed with a dual wave insulin bolus. This study evaluated the effect of a simple bolus on glycemia following consumption of traditionally prepared pizzas with long (22 hours) or short (8 hours) dough fermentation periods.

DETAILED DESCRIPTION:
All participants received pizza prepared in one of two ways, as described below, on two separate days. On the first day, they were given a pizza prepared with dough fermented for 8 hours (pizza A), and on the second study day they received a pizza prepared with dough fermented for 24 hours (pizza B). Participants and their parents were blinded to the type of pizza served on each day. Both meals were served at 7.00 pm at the pizzeria where the pizza had been prepared, and consumed within 30 minutes.

Children and adolescents aged between 4 and 18 years with type 1 diabetes were eligible for inclusion in the study if they had received SIP therapy (MiniMed™ 640G, Medtronic, Tolochenaz, Switzerland) for at least 3 months One pizza of each type was prepared for chemical analysis

ELIGIBILITY:
Inclusion Criteria:

* type 1 diabetes if they had received sensor integrated pump (SIP) therapy for at least 3 months

Exclusion Criteria:

* Patients with HbA1c >8.5% (69 mmol/mol), celiac disease, other food allergies or concurrent illness

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 38 (Actual)
Dates: Start 2018-02-14 (Actual); Primary Completion 2018-03-21 (Actual); Study Completion 2018-10-01 (Actual)

PRIMARY OUTCOMES:
Continuous glucose sensor data | 11 hours
  mmol/L

SECONDARY OUTCOMES:
Content of carbohydrates | 1 hour
  µg/g

OTHER OUTCOMES:
Content of amino acids | 1 hour
  µg/g

CONTACTS AND LOCATIONS:
Locations (1):
- Centro di Diabetologia Pediatrica "G.Stoppoloni", Naples, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Combet E, Jarlot A, Aidoo KE, Lean ME. Development of a nutritionally balanced pizza as a functional meal designed to meet published dietary guidelines. Public Health Nutr. 2014 Nov;17(11):2577-86. doi: 10.1017/S1368980013002814. Epub 2013 Oct 28. PMID 24160252
- [Result] Gallus S, Tavani A, La Vecchia C. Pizza and risk of acute myocardial infarction. Eur J Clin Nutr. 2004 Nov;58(11):1543-6. doi: 10.1038/sj.ejcn.1601997. PMID 15138460
- [Result] Ahern JA, Gatcomb PM, Held NA, Petit WA Jr, Tamborlane WV. Exaggerated hyperglycemia after a pizza meal in well-controlled diabetes. Diabetes Care. 1993 Apr;16(4):578-80. doi: 10.2337/diacare.16.4.578. PMID 8462382
- [Result] Mauseth R, Lord SM, Hirsch IB, Kircher RC, Matheson DP, Greenbaum CJ. Stress Testing of an Artificial Pancreas System With Pizza and Exercise Leads to Improvements in the System's Fuzzy Logic Controller. J Diabetes Sci Technol. 2015 Sep 14;9(6):1253-9. doi: 10.1177/1932296815602098. PMID 26370244
- [Result] Pankowska E, Blazik M, Groele L. Does the fat-protein meal increase postprandial glucose level in type 1 diabetes patients on insulin pump: the conclusion of a randomized study. Diabetes Technol Ther. 2012 Jan;14(1):16-22. doi: 10.1089/dia.2011.0083. Epub 2011 Oct 20. PMID 22013887
- [Result] De Palma A, Giani E, Iafusco D, Bosetti A, Macedoni M, Gazzarri A, Spiri D, Scaramuzza AE, Zuccotti GV. Lowering postprandial glycemia in children with type 1 diabetes after Italian pizza "margherita" (TyBoDi2 Study). Diabetes Technol Ther. 2011 Apr;13(4):483-7. doi: 10.1089/dia.2010.0163. Epub 2011 Feb 28. PMID 21355715
- [Result] Jones SM, Quarry JL, Caldwell-McMillan M, Mauger DT, Gabbay RA. Optimal insulin pump dosing and postprandial glycemia following a pizza meal using the continuous glucose monitoring system. Diabetes Technol Ther. 2005 Apr;7(2):233-40. doi: 10.1089/dia.2005.7.233. PMID 15857224
- [Derived] Zanfardino A, Confetto S, Curto S, Cocca A, Rollato AS, Zanfardino F, Troise AD, Testa V, Bologna O, Stanco M, Piscopo A, Cohen O, Miraglia Del Giudice E, Vitaglione P, Iafusco D. Demystifying the Pizza Bolus: The Effect of Dough Fermentation on Glycemic Response-A Sensor-Augmented Pump Intervention Trial in Children with Type 1 Diabetes Mellitus. Diabetes Technol Ther. 2019 Dec;21(12):721-726. doi: 10.1089/dia.2019.0191. Epub 2019 Aug 8. PMID 31335171